CLINICAL TRIAL: NCT01548768
Title: RHYTHM (RHeumatoid Arthritis studY of THe Myocardium): How Rheumatoid Arthritis (RA) and Tumor Necrosis Factor (TNF) Inhibitors Affect the Myocardial Structure and Function.
Brief Title: RHYTHM (Formerly Escape II Myocardium)
Acronym: RHYTHM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Joan M. Bathon, Professor Medicine, Rheumatology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAI1026; 7R01AR050026-07 (NIH)
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Cardiovascular disease; Myocardium; TNF-alpha inhibitors; ESCAPE; Co-morbidities; RHYTHM
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases | interventions — Tumor Necrosis Factor Inhibitors; Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients - DMARDs + TNF Inhibitors (Experimental): Patients will receive a TNF inhibitor in addition to their current treatment in an open label protocol for increased disease activity and in the context of standard of care.
  Interventions: Drug: TNF inhibitors; Drug: DMARDs
- Patients - DMARDs only (Active Comparator): Patients will receive their current treatment in an open label protocol in the context of standard of care.
  Interventions: Drug: DMARDs
- Healthy Volunteers (No Intervention): Subjects without RA who will function as controls.

INTERVENTIONS:
Drug: TNF inhibitors — TNF inhibitors are an FDA approved class of medications indicated for the treatment of RA when initial treatment (usually with methotrexate) has failed to achieve remission of RA disease activity. TNF inhibitors are part of the standard of care management of RA.
  The possible TNF inhibitors are: Remicade, Humira, Enbrel, Cimzia, Simponi.
  Other Names: Anti-TNF drugs
  Arms: Patients - DMARDs + TNF Inhibitors
Drug: DMARDs — Standard of care treatment for RA, such as Methotrexate or other disease-modifying antirheumatic drugs.
  Other Names: Disease-modifying antirheumatic drugs
  Arms: Patients - DMARDs + TNF Inhibitors; Patients - DMARDs only

SUMMARY:
For aim 1, the proposed studies will be performed in 150 patients with RA and 25 subjects without RA (healthy volunteers) who will function as controls.

For aim 2, 25 of the patients enrolled in aim 1 (who are in need for further treatment due to increased RA activity despite their current treatment) will be recruited to continue in the study for an additional 24 (+/- 2) weeks (or 6 months). These patient will receive a TNF inhibitor in addition to their current treatment in an open label protocol for increased disease activity and in the context of standard of care.

The investigators hypothesize that anti-TNF agents in RA patients without heart disease will not adversely affect the heart (will not cause a detrimental change in heart structure or its function).

DETAILED DESCRIPTION:
Patients with Rheumatoid Arthritis (RA) have a shortened life expectancy compared to the general population. Cardiovascular disease (CVD), including heart failure (HF), is the primary cause of the extra deaths in RA. HF, in general, results from failure of the heart muscle to pump adequately. In other words the heart muscle in HF becomes "weak". In patients without RA, the heart muscle gets larger before symptoms of HF appear. Contrary to that, patients with RA have reduced heart size and reduced heart strength. This may mean that in RA the pathway to heart failure may be different compared to what happens in patients without RA. It is possible - for example - that in RA the heart muscle becomes smaller before it becomes weak (while in non-RA patients the heart muscle becomes larger before it becomes weak). It is possible that cells that create inflammation in the joints may also do the same in the heart muscle making it smaller, thinner and eventually weaker.

Patients with RA nowadays can be treated with a variety of medications for their joint inflammation. These medications are powerful and have reduced the risk of permanent joint damage and disability. However it is unknown what is the effect of these medications on the heart size and strength and whether they increase or decrease the risk for cardiovascular disease and heart failure.

Among the medications used for RA are medications called TNF inhibitors. They are usually prescribed to patients who have joint inflammation that has not responded to treatment with the first line medication Methotrexate. Data in non-RA patients with advanced heart failure suggest that anti-TNF agents may not help heart failure and may even be harmful. However, the effect of these agents on the hearts of RA patients has never been directly studied. Some observational studies suggest that RA patients treated with TNF inhibitors have a lower risk of developing heart disease. Overall the knowledge regarding the effect of TNF inhibitors on RA patients heart function is limited.

ELIGIBILITY:
For RA patients (150 patients):

INCLUSION CRITERIA

* Diagnosis of Rheumatoid Arthritis by 2010 American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) diagnostic criteria
* Age>18 years old
* Moderate to high RA disease activity defined by a Clinical Disease Activity Index (CDAI) of >10
* Stable dose of Methotrexate for 6 weeks prior to enrollment
* Stable doses of Nonsteroidal anti-inflammatory drug (NSAID) and prednisone (if already taking these medications) for 2 weeks prior to study

EXCLUSION CRITERIA

* Prior self reported or physician diagnosed CV event (MI; angina; stroke or Transient Ischemic Attach (TIA); Heart Failure (HF); prior CV procedure (e.g., coronary artery bypass graft, angioplasty, valve replacement, pacemaker)
* Contraindications to having a PET-CT scan or receive adenosine or Fludeoxyglucose (FDG)
* Active treatment for Cancer
* Uncontrolled hypertension
* Diabetes
* Smoking
* Treatment with a TNF inhibitor or other biologic currently or within the last 6 months
* Current treatment with "Triple Therapy" or within the last 2 months
* Untreated positive purified protein derivative (PPD) tuberculosis skin test or active tuberculosis
* History of Lymphoma and Melanoma
* Ejection Fraction (EF) < 40% (if not known in advance then the Study Visit I Echocardiogram results will be used to exclude the patient from randomization and follow up)
* Change in NSAID/Prednisone dosage in last 2 weeks
* Participation in other research studies involving imaging/radiation exposure

For non-RA subjects (25 controls):

INCLUSION CRITERIA

* Age>18 years old
* Absence of diagnosis of RA

EXCLUSION CRITERIA

* Prior self reported or physician diagnosed CV event (MI; angina; stroke or Transient Ischemic Attach (TIA); Heart Failure (HF); prior CV procedure (e.g., coronary artery bypass graft, angioplasty, valve replacement, pacemaker)
* Contraindications to having a PET-CT scan or receive adenosine or FDG
* Uncontrolled hypertension
* Participation in other research studies involving imaging/radiation exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-10-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Bathon, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amigues I, Tugcu A, Russo C, Giles JT, Morgenstein R, Zartoshti A, Schulze C, Flores R, Bokhari S, Bathon JM. Myocardial Inflammation, Measured Using 18-Fluorodeoxyglucose Positron Emission Tomography With Computed Tomography, Is Associated With Disease Activity in Rheumatoid Arthritis. Arthritis Rheumatol. 2019 Apr;71(4):496-506. doi: 10.1002/art.40771. Epub 2019 Feb 28. PMID 30407745
- See also: Click here for information about this study — http://www.rheumatologyatcolumbia.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients - DMARDs + TNF Inhibitors: Patients will receive a TNF inhibitor in addition to their current treatment in an open label protocol for increased disease activity and in the context of standard of care.
  TNF inhibitors: TNF inhibitors are an FDA approved class of medications indicated for the treatment of RA when initial treatment (usually with methotrexate) has failed to achieve remission of RA disease activity. TNF inhibitors are part of the standard of care management of RA.
  The possible TNF inhibitors are: Remicade, Humira, Enbrel, Cimzia, Simponi.
  DMARDs: Standard of care treatment for RA, such as Methotrexate or other disease-modifying antirheumatic drugs.
- Patients - Cross Sectional (RA): A cohort of patients with Rheumatoid Arthritis will undergo the baseline study visit only (no randomization to treatment). Note, that those who were randomized, their data will be utilized in the full cross sectional analysis.
Period: Overall Study
Arm/Group | Patients - DMARDs + TNF Inhibitors | Patients - DMARDs Only | Healthy Volunteers | Patients - Cross Sectional (RA)
Started | 8 | 4 | 16 | 121
Completed | 7 | 2 | 15 | 117
Not Completed | 1 | 2 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Non-Compliance | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: RA participants=133, Healthy Volunteers=16
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients - DMARDs + TNF Inhibitors | Patients - DMARDs Only | Healthy Volunteers | Patients - Cross Sectional (RA) | Total
Number analyzed (Participants) | 8 | 4 | 16 | 121 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 15 | 105 | 130
  >=65 years | 0 | 2 | 1 | 16 | 19
Age, Continuous [Mean (Full Range); unit: years] | 55.125 [32 to 64] | 56 [26 to 70] | 52 [28 to 68] | 55.6 [23 to 80] | 54.38 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 12 | 105 | 127
  Male | 2 | 0 | 4 | 16 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4 | 52 | 60
  Not Hispanic or Latino | 5 | 3 | 12 | 69 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 5 | 28 | 36
  White | 5 | 3 | 11 | 53 | 72
  More than one race | 0 | 0 | 0 | 36 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Myocardial FDG Uptake
Description: This is designed to evaluate the baseline characteristics of the cross sectional RA cohort to understand the correlation of disease activity measured by the Clinical Disease Activity Index (CDAI) with myocardial inflammation measured by fluorodeoxyglucose (FDG) uptake in positron emission tomography (PET) scan at the baseline visit. Myocardial FDG uptake is classified as "diffuse" or "focal."
Time Frame: Baseline
Population: 2 RA patients and 1 healthy volunteer (control subject) were not included in this analysis population because the subjects withdrew study participation prior to scan (no data were collected).
Measure: Count of Participants; unit: Participants
Groups:
- Patients - Cross Sectional (RA): A cohort of patients with Rheumatoid Arthritis who underwent the baseline visit analysis and completed the visit in the full cross sectional analysis.
- Healthy Volunteers: A cohort of healthy volunteers (those without an autoimmune or history of cardiac illness) was utilized. n=16 were recruited directly, while n=11 were recruited via the CUIMC Nuclear Cardiology archive.
Arm/Group | Patients - Cross Sectional (RA) | Healthy Volunteers
Number analyzed (Participants) | 119 | 15
Participants
  Diffuse FDG Uptake | 21 | 4
  Focal FDG Uptake | 25 | 1
  No FDG Uptake | 73 | 10

2. Secondary Outcome: Number of Participants With Myocardial FDG Uptake After Escalation of RA Pharmacotherapy
Description: This is designed to measure the myocardial inflammation, and its association with change in CDAI, after ramp-up of RA therapy over 6 months. Measurements are taken at baseline and 6-months post treatment escalation. Myocardial FDG uptake is classified as "diffuse" or "focal."
Time Frame: Baseline, 6-Month Follow-up
Population: 2 TNFi, and 2 DMARDs and 1 healthy volunteer (control subject) were not included in this analysis population because the subjects withdrew participation prior to study completion or scan (no data were collected).
Measure: Number; unit: participants
Groups:
- RA Patients - Pharmacotherapy Escalation (TNFi): Participants were randomized to TNFi or DMARD therapy.
  Patients will receive their current treatment in an open label protocol in the context of standard of care.
  TNFi: biologic treatment for RA, such as Humira, Enbrel, Remicade,
- RA Patients - Pharmacotherapy Escalation (DMARD): Participants were randomized to TNFi or DMARD therapy.
  Patients will receive their current treatment in an open label protocol in the context of standard of care.
  DMARDs: Standard of care treatment for RA, such as Methotrexate or other disease-modifying antirheumatic drugs.
Arm/Group | RA Patients - Pharmacotherapy Escalation (TNFi) | RA Patients - Pharmacotherapy Escalation (DMARD) | Healthy Volunteers
Number analyzed (Participants) | 6 | 2 | 15
participants
  Focal Baseline FDG Uptake | 1 | 1 | 1
  Focal Follow-up FDG Uptake | 1 | 0 | NA — Healthy Controls were not re-scanned 6-months later, and served as a comparison marker
  Diffuse Baseline FDG Uptake | 4 | 1 | 4
  Diffuse Follow-up FDG Uptake | 2 | 0 | NA — Healthy Controls were not re-scanned 6-months later, and served as a comparison marker

3. Secondary Outcome: LV Structure (Mean EDVI) in Association With Myocardial FDG Uptake
Description: This is designed to evaluate the baseline characteristics of the entire RA cohort to understand the association of myocardial inflammation measure by FDG uptake with measures of left ventricular (LV) structure measured by 2D/3D echocardiogram at the baseline visit.
Time Frame: Baseline
Population: Only 119 out of 121 subjects had data analyzed due to 2 subject withdrawals prior to scan.
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Patients - Cross Sectional (RA) | Healthy Volunteers
Number analyzed (Participants) | 119 | 16
ml/m^2 | 53.8 (11) | 49.1 (12.9)

4. Secondary Outcome: LV Function (Mean Stroke Volume Index) in Association With Myocardial FDG Uptake
Description: This is designed to evaluate the baseline characteristics of the entire RA cohort to understand the association of myocardial inflammation measure by FDG uptake with measures of left ventricular (LV) function measured by 2D/3D echocardiogram at the baseline visit.
Time Frame: Baseline
Population: Only 119 out of 121 subjects had data analyzed due to 2 subject withdrawals prior to scan.
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Patients - Cross Sectional (RA) | Healthy Volunteers
Number analyzed (Participants) | 119 | 16
ml/m^2 | 58.6 (13.9) | 31.3 (7.5)

ADVERSE EVENTS:
Time Frame: For those who underwent the baseline scans only (RA cross-sectional cohort, Healthy Controls), the gathering of adverse events were determined from the events from the visit alone (either acute, or patient-reported follow-up); For the group escalated in treatment therapy (n=12), adverse events were collected from baseline visit/randomization to the end-of-study safety visit conducted 6-8 weeks after the 6-month study visit.
Description: An adverse event (AE) is any undesirable sign, symptom or medical condition occurring after starting study drug (or therapy). Medical conditions/diseases present before starting study treatment are only considered adverse events if they worsen after starting study therapy. In addition all adverse events regardless of whether they constitute unanticipated problems as well as AEs thought to be possibly related to study procedures will also be reported to IRB, safety officer, SMC, and NIH/NIAMS.
Arm/Group | RA Patients - Pharmacotherapy Escalation (TNFi) | RA Patients - Pharmacotherapy Escalation (DMARD) | Healthy Volunteers | Patients - Cross Sectional (RA)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/16 | 0/121
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/4 | 0/16 | 0/121
Other Adverse Events (participants affected / at risk) | 1/8 | 0/4 | 0/16 | 6/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA Patients - Pharmacotherapy Escalation (TNFi) (N=8) | RA Patients - Pharmacotherapy Escalation (DMARD) (N=4) | Healthy Volunteers (N=16) | Patients - Cross Sectional (RA) (N=121)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant was admitted during overseas travel to hospital in Ecuador for an episode of acute dyspnea - she spent one night in a hospital in Panama before returning to the US.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA Patients - Pharmacotherapy Escalation (TNFi) (N=8) | RA Patients - Pharmacotherapy Escalation (DMARD) (N=4) | Healthy Volunteers (N=16) | Patients - Cross Sectional (RA) (N=121)
Worsening Migraine (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject w/ h/o migraine; during study visit, mild migraine in morning worsened (BP 140/69, HR 100) - given acetaminophen 500mg x2 - decision made to admit to ED for observation. Same-day discharge from ED.
Mobitz II Heart Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Could not tolerate adenosine - subject went into heart block (otherwise asymptomatic); IRB gave approval for regadenoson on re-try later.
Angina (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Angina during adenosine stress test w/ ischemic ECG changes during test. Resolved on completion of test.
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Short run of atrial tachycardia which self-reverted to normal sinus rhythm after 100mg aminophyllin. No re-occurance.
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject had panic attack during stress scan - test was aborted and not retried.
Thrombophlebitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject had swelling from IV site; prescribed Keflex for 10 days, which resolved.
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject reported new pruritic skin rash (c/w eczema on exam) on start of study medication. Study medication d/c'ed 1mnth later and initiated medrol w/ good response. Later followed up with dermatology who confirmed eczema.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT01548768/Prot_SAP_000.pdf